CLINICAL TRIAL: NCT03965104
Title: Improving Hypertension Detection and Control Through a Hypertension Certification Program Based Upon the Hypertension Canada Guidelines (RxPATH)
Brief Title: Improving Hypertension Detection and Control Through a Hypertension Certification Program Based Upon the Hypertension Canada Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Hypertension Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00090012
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial with the unit of randomization being the pharmacy
Who Masked: Participant
Masking Description: By necessity, pharmacists in the intervention groups cannot be blinded. However, pharmacists will not be told about the cluster randomization, just that they will be contacted about when they will receive the HC-PCP. During the control period, pharmacists will be told that their patients will be enrolled in an observational hypertension registry to prepare for the intervention phase.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention pharmacists (Experimental): Will receive the HC-PCP prior to starting enrollment, and then will provide care to their patients, which will include risk assessment, prescribing of antihypertensive medications, and follow-up monthly according to the Hypertension Canada Guidelines.
  Interventions: Behavioral: Hypertension Canada Professional Certification Program: HC-PCP
- Control pharmacists (No Intervention): Will provide usual pharmacist care. All patients with blood pressure above target will be entered into the study database and serve as the control group. No specific interventions or follow-up will be mandated other than usual pharmacist care, although all patients will be assessed at 3 months to determine change in BP since enrollment (the primary outcome).

INTERVENTIONS:
Behavioral: Hypertension Canada Professional Certification Program: HC-PCP — The HC-PCP is a certification program which aims to provide training to generalist primary care providers in the screening, prevention, and management of hypertension.The competencies assessed in the program have been validated for their importance through a national survey of hypertension experts and primary care providers.
  Arms: Intervention pharmacists

SUMMARY:
This study will assess the impact of a hypertension management certification program for community pharmacists on the blood pressure control of patients managed by the pharmacists enrolled. The investigators will compare the systolic blood pressure of patients identified to have hypertension in the community that are followed by pharmacists who have undergone the certification course, and compare their blood pressure outcomes to subjects managed by pharmacists who have not yet received the training.

DETAILED DESCRIPTION:
Hypertension Canada proposes the first "Hypertension Canada Professional Certification Program"(HC-PCP), specifically designed for Alberta pharmacists, to provide care and support to those at risk for or living with hypertension. Through this program, the investigators hope to help with prevention of the costly and chronic conditions to which hypertension often leads, like kidney failure, stroke, and heart disease.

The HC-PCP aims to provide training to pharmacists in the screening, prevention, and management of hypertension. It has been identified that the development and implementation of this certification program provides a unique opportunity to evaluate the impact of such a program on blood pressure reduction.

The investigators are aiming to assess the impact of pharmacist management on blood pressure control in patients with hypertension.

The development of the HC-PCP and the evaluation of its impact will occur in 2 phases. Phase 1 involves the development and implementation of the educational portion of the certification program. Phase 2 involves conducting a 1 year long study to assess the impact of the HC-PCP on blood pressure in patients with poorly controlled hypertension. This will be launched in pharmacies in Alberta.

ELIGIBILITY:
Inclusion Criteria:

* Patients with poorly controlled blood pressure (>140/90mmHg or >130/80mmHg if they have diabetes).

Exclusion Criteria:

* Unwilling to sign the consent form.
* Unwilling to participate in follow up visits.
* Current hypertension urgency or emergency (SBP > 180mmHg or DBP > 120mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
The difference in change in systolic blood pressure between Intervention and Control patients. | From baseline to 3 month follow-up, and up to one year
  To detect a 7 millimeters of mercury (mmHg) or greater difference in systolic blood pressure.

SECONDARY OUTCOMES:
Consultant Satisfaction Questionnaire | 6 months following follow up
  patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, PharmD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No